CLINICAL TRIAL: NCT02479685
Title: Prospective Randomized Trial on Laparoscopic Subtotal Hysterectomy During Sacral Colpopexy for the Treatment of Severe Pelvic Organ Prolapse (POP) With Bipolar Laparoscopic Loop/Bipolar Morcellator vs Conventional Monopolar Hook/Conventional Morcellator
Brief Title: SORD-BILL Vs Conventional Options During Sacral Colpopexy for POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Giuseppe Campagna (Unknown); Cristiano Rossitto (Unknown); Andrea Morciano (Unknown)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SORD-BILL
Record Dates: First submitted 2015-01-05; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SORD-BILL (Experimental): PKS BILL: bipolar laparoscopic loop (a laparoscopic loop using advanced bipolar energy) (Olympus Medical Systems Corp, Tokyo) and PKS PlasmaSORD (Solid Organ Removal Device) for subtotal hysterectomy and uterine morcellation, respectivelly, during sacral colpopexy for Pelvic Organ Prolapse.
  Interventions: Procedure: PKS BILL-PKS PlasmaSORD Versus Conventional surgical techniques
- STANDARD (Active Comparator): Conventional monopolar hook and conventional mechanic morcellator for subtotal hysterectomy and uterine morcellation, respectivelly, during sacral colpopexy for Pelvic Organ Prolapse.
  Interventions: Procedure: PKS BILL-PKS PlasmaSORD Versus Conventional surgical techniques

INTERVENTIONS:
Procedure: PKS BILL-PKS PlasmaSORD Versus Conventional surgical techniques — To verify if the operative time of a standard laparoscopic sacral colpopexy associated to subtotal hysterectomy for the treatment of POP could be further reduced using PKS BILL: bipolar laparoscopic loop (a laparoscopic loop using advanced bipolar energy) (Olympus Medical Systems Corp, Tokyo) and PKS PlasmaSORD (Solid Organ Removal Device) vs. conventional monopolar hook and conventional mechanic morcellator.

SUMMARY:
This prospective randomized pilot study is aimed to verify if the operative time of a standard laparoscopic sacral colpopexy associated to subtotal hysterectomy for the treatment of POP could be further reduced using PKS BILL: bipolar laparoscopic loop (a laparoscopic loop using advanced bipolar energy) (Olympus Medical Systems Corp, Tokyo) and PKS PlasmaSORD (Solid Organ Removal Device) vs. conventional monopolar hook and conventional mechanic morcellator.

DETAILED DESCRIPTION:
Introduction Pelvic-organ prolapse, in which the pelvic organs (uterus, bladder, and bowel) protrude into or past the vaginal introitus, is a condition often treated with surgery1,2. Women have an 11 percent risk of surgery for prolapse or urinary incontinence by 80 years of age, and of this 11 percent, almost one third of the women have a second surgery3. This fact points to the need for improved treatment of pelvic-floor disorders. Numerous surgical procedures have been described for the management of POP. Vaginal surgery may be associated with less postoperative pain and a more rapid return to daily living than abdominal repair4,5. However, in a randomised study, sacrocolpopexy was twice as likely to result in optimal anatomical outcome as vaginal surgery6. Laparoscopic sacrocolpopexy provides the potential to combine the success rates of an abdominal approach with the faster recovery associated with a minimally invasive technique. Tissue dissection and mesh placement may also be facilitated by the magnification and field of view permitted by the laparoscopic approach7-10. These benefits must be balanced against a longer operating time from 150 to 250 minutes according to surgeons' experience. In addition, this procedure is often associated to subtotal hysterectomy (LSH) for the reasons of prevention (post-menopause age) or uterine diseases, which improve still more the operating time. Literature studies reports that the use of electrosurgical loop decreased the time required for resection of the uterine cervix during LSH for benign uterine conditions. Moreover LSH can be performed more easily with a powered morcellator for removal of the uterus. These devices facilitate and increase the safety of this procedure11,12.

However, the available laparoscopic morcellators may be difficult to use (weight, ergonomics, etc.) and there are potentially serious complications unreported in the medical literature13.

This prospective randomized pilot study is aimed to verify if the operative time of a standard laparoscopic sacral colpopexy associated to subtotal hysterectomy for the treatment of POP could be further reduced using PKS BILL: bipolar laparoscopic loop (a laparoscopic loop using advanced bipolar energy) (Olympus Medical Systems Corp, Tokyo) and PKS PlasmaSORD (Solid Organ Removal Device) vs. conventional monopolar hook and conventional mechanic morcellator.

Secondary endopoints of this comparison are incidence of intra- or postoperative complications estimated blood loss, postoperative pain (evaluated by VAS), days of hospitalization and costs for the health care system.

Statistical Analysis and Study Design This is a single Institution prospective randomized clinical trial conducted at the Catholic University of the Sacred Heart, Rome.

To have an imbalanced results and to reduce any bias, a randomization list has been checked.

Probability (p) values will be considered to be statistically significant at the <0.05 level.

There will be recruited 50 patients to treat using PK BiLL/PKS plasmasord and 50 patients to treat with standard monopolar hook/standard morcellator comparing these two techniques in terms of operative time, estimated blood loss and other intra- or post operative complications, postoperative pain, days of hospitalization, costs. All patients will be adequately informed and inserted in the study only after having read and signed an informed consent. Diagnostic, clinical and surgical data of each patient will be prospectively recorded. At the end of the procedure, a schedule will be compiled with intraoperative data. All clinical and histologic data will be recorded prospectively using a database. Pain associated with the procedure will be evaluated by a subjective assessment (analysis of VAS scale values reported by patients at 8 and 24 hours after surgery). Post-operative complications will be evaluated during the first 30 days after surgery according to Dindo's classification14.

Consort diagram of the study

Study Objectives

Primary endpoint To compare operative time for laparoscopic sacral colpopexy associated to subtotal hysterectomy for the treatment of POP using PKS BILL and PKS plasmasord technology (bipolar laparoscopic loop and bipolar morcellator) vs. conventional monopolar hook and conventional mechanic morcellator in order to reduce this operative time.

Secondary endpoints To compare

* Intra- or post operative complications (Urinary, Intestinal, Nervous)
* Estimated blood loss
* Postoperative pain
* Days of hospitalization
* Costs for the health care system.

Inclusion/exclusion criteria

For patients

* Age ≤ 80 years
* Patient's informed consent
* American Society of Anesthesiologists: < class III or IV
* Physiologic, surgical or iatrogenic menopause.
* No previous major abdominal surgical procedures

For diseases

* POP-Q stage III/IV for anterior and/or apical compartment; stage <III for posterior compartment.
* No uterine cervix dysplasia or endometrial disorders.
* No uterine size larger than conform 10 weeks gestation

Study procedures Standard sacral colpopexy with subtotal hysterectomy With the patient in the Trendelenburg position (≥30°), after insertion of a 16F Foley urethral catheter, adequate pneumoperitoneum was induced. Uterine manipulator is used to move the uterus.A 10-mm laparoscope was introduced through the umbilicus and two 5-mm trocars were placed 2 cm medially and superiorly to the anterosuperior iliac spines. After thorough evaluation of the peritoneal cavity and, if necessary, completion of adhesiolysis, an additional 5- to 12-mm trocar was placed under visual control in the midline half way between the pubic symphysis and umbilicus. In the case of obesity or short umbilicopubic length, the 5-to 12-mm trocar was placed at the umbilicus and the 10-mm optical trocar was inserted in midline half way between the xiphoid process and umbilicus. The first step of LSC consisted of locating useful anatomic landmarks (outline of the promontory, iliac bifurcation, left common iliac vein, right ureter) and exposing the longitudinal vertebral ligament covering the sacral promontory. This was accomplished by opening the parietal peritoneum and gentle sharp and blunt dissection of retroperitonal tissue. Median sacral vessels were pushed back inward during dissection or coagulated if necessary. Then the peritoneal incision was prolonged along the right pelvic wall up to the uterine isthmus, paying careful attention to the ureter when mesh subperitonealization was scheduled.

The subtotal hysterectomy started now. The round ligaments are coagulated and cut to enter the retroperitoneum. The broad ligaments/ovarian pedicles are sealed with bipolar diathermy and divided with monopolar scissors. Anterior and posteriors leaves of the broad ligaments peritoneum are divided with monopolar scissors. The incision is carried anteriorly. The bladder peritoneum is incised distal to the cervicouterine junction. Paravescical and pararectal spaces are developed. After both uterine arteries were coagulated using bipolar diathermy and monopolar forceps and the bladder dissection was completed, supracervical separation of the uterus wasperformed using a monopolar hook after removal of the uterine manipulator. The uterus was then morcellated by drawing the specimen into the morcellator (ROTOCUT G1 Morcellator, KARL STORZ GmbH & Co. KG, Tuttlingen, Germany).

The pouch of Douglas was incised between the left and right uterosacral ligaments and the rectovaginal space was dissected along the posterior vaginal wall. Margins of dissection were the perineal body inferiorly and rectovaginal ligament laterally. To cover all the dissection space without tension, an adequately shaped Prolene mesh (Ethicon, Inc) was placed and fixed to the vaginal wall by five 3-0 nonabsorbable sutures. The first suture was applied in midline at the perineal apex of the mesh. Two sutures for each side were applied on the middle and upper portions of the posterolateral vaginal walls. The vesicouterine peritoneum was opened and vesicouterine and vesicovaginal spaces were dissected along the uterine and vaginal walls. Dissection limits were the trigonal region (emphasized by the Foley catheter) inferiorly and bladder pillars laterally. Also in this case an adequately shaped Prolene mesh covering all the dissection space without tension was inserted and fixed to the vaginal wall with five 3-0 nonabsorbable sutures. The first suture was applied at midline at the vesical apex of the mesh. Two sutures for each side were located on the middle and upper portions of anterolateral vaginal walls. The peritoneum of the right broad ligament between the round ligament-ovarian ligament superiorly and parametrial portion of uterine vessels inferiorly was incised so as to rejoin the previous right peritoneal incision, and the anterior mesh was passed through the incision. The two meshes were threaded up toward the promontory under visual control from the vagina so as to lift the prolapse vaginal walls without excessive tension. Meshes were fixed to the longitudinal vertebral ligament with one 0 non-absorbable suture on a noncutting needle . The operation was completed by re-peritonealization.

PKS BiLL technology Using PKS bipolar laparoscopic loop can simplify cervical amputation and decreased the time required for the detachment of the uterine corpus, which many consider the more difficult part of laparoscopic subtotal hysterectomy. In addition, the loop system allows the supracervical separation of the uterus at or above the level of the coagulated uterine vessels, therefore minimising the risk of slippage or retraction of the vessels. The bipolar technology could add an ulterior advantage in terms of safety and operating procedure time reduction.

In the same way the use of PKS plasmasord bipolar morcellator could reduce the risk of injuries. The lightness of this instrument could increase the procedure feasibility.

ELIGIBILITY:
Inclusion Criteria:

For patients

* Age ≤ 80 years
* Patient's informed consent
* American Society of Anesthesiologists: < class III or IV
* Physiologic, surgical or iatrogenic menopause.
* No previous major abdominal surgical procedures

For diseases

* POP-Q stage III/IV for anterior and/or apical compartment; stage <III for posterior compartment.
* No uterine cervix dysplasia or endometrial disorders.
* No uterine size larger than conform 10 weeks gestation

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Operative time for LPS subtotal hysterectomy and sacral colpopexy | participants will be followed for the duration of hospital stay, , an expected average of 5 weeks
  operative time will be calculated from the entrance in the abdominal cavity to the closure of the skin trocar accesses

SECONDARY OUTCOMES:
incidence of intra- or postoperative complications estimated (blood loss, postoperative pain (evaluated by VAS), days of hospitalization and costs for the health care system). | participants will be followed for the duration of hospital stay, , an expected average of 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Professor, Principal Investigator — Catholic University of the Sacred Heart - Rome
Locations (1):
- Catholic University of Sacred Heart Rome,, Rome, Rome, Italy

REFERENCES:
- [Derived] Campagna G, Morciano A, Rossitto C, Panico G, Naldini A, Ercoli A, Cervigni M, Scambia G. A new approach to supracervical hysterectomy during laparoscopic sacral colpopexy for pelvic organ prolapse: A randomized clinical trial. Neurourol Urodyn. 2017 Mar;36(3):798-802. doi: 10.1002/nau.23030. Epub 2016 Apr 29. PMID 27128776